CLINICAL TRIAL: NCT00312819
Title: Randomized Phase 2 Trial of Treatment of Advanced Non Small Cell Lung Carcinoma With/Without Disulfiram and Cisplatin Navelbine
Brief Title: Initial Assessment of the Effect of the Addition of Disulfiram (Antabuse) to Standard Chemotherapy in Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Augusta Hospital, Berlin (Other)
Responsible Party: hovav nechushtan, HadassahHMO
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DVC1.03-HMO-CTIL
Record Dates: First submitted 2006-04-10; First posted 2006-04-11 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2009-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cel lung cancer; chemotherapy; randomized phaseII; disulfiram; antiangiogenesis; placebo
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: chemotherapy +/- disulfiram

SUMMARY:
Recent studies in laboratory animals demonstrate the ability of disulfiram to significantly inhibit the growth and metastasis of a mouse model of lung cancer. Work with cells in vitro support the idea that this inhibition is mainly due to the inhibition of angiogenesis - the formation of new blood vessels in the tumor. Furthermore, it was found out that the best effect has been obtained when disulfiram has been used not at the highest dose but at an optimal dose, which is smaller. Thus, this trial will assess the addition of disulfiram to chemotherapy in non-small cell lung cancer (NSCLCA).

DETAILED DESCRIPTION:
Metastatic non small cell lung cancer remains a deadly disease with median survival times of several months. Any treatment which can prolong patients' survival without causing severe side effects is of course an important addition to our limited arsenal in the fight against this disease. A recent article by Marikowsky and colleagues extended significantly our knowledge regarding the possible activity of disulfiram (well known in its commercial name Antabuse) as an anticancer agent (Marikowsky et al Int J of cancer 97 :34 2002). In this article it was demonstrated that disulfiram has potent antitumor activity and that it can act as a significant inhbitor of angiogenesis.

Since disulfiram has been well tolerated by thousands of patients, and there are observations that anti angiogenic therapy enhances the effect of chemotherapy (for example bevacizumab in combination with chemotherapy in colon carcinoma) we decided to conduct a clinical trial assessing the effect of the addition of this drug at moderate doses to chemotherapy which is used as one of the standard therapies in lung cancer. In order to obtain information regarding the effect of the addition of this drug, only 50% of the patients will be treated with the drug and the rest will be treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic non-small cell lung cancer
* Previously untreated
* ECOG performance status (PS) 0-1
* Liver function tests within the norm

Exclusion Criteria:

* Over 18
* Willingness to abstain from alcohol
* Not pregnant
* Without a psychiatric history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
tumor response disease free survival survival | 3 years

SECONDARY OUTCOMES:
Clinical response
treatment tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Hovav Nechushtan, MD, PhD, Principal Investigator — Hadassah Medical Center Ein Kerem; Nili Peylan-Ramu, MD, Study Chair — Hadassah Ein Kerem Medical Center; Maya Gotfrid, MD, Study Chair — Meir Medical Center Kfar Saba
Locations (1):
- Oncology Institute Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Marikovsky M, Nevo N, Vadai E, Harris-Cerruti C. Cu/Zn superoxide dismutase plays a role in angiogenesis. Int J Cancer. 2002 Jan 1;97(1):34-41. doi: 10.1002/ijc.1565. PMID 11774241
- [Derived] Nechushtan H, Hamamreh Y, Nidal S, Gotfried M, Baron A, Shalev YI, Nisman B, Peretz T, Peylan-Ramu N. A phase IIb trial assessing the addition of disulfiram to chemotherapy for the treatment of metastatic non-small cell lung cancer. Oncologist. 2015 Apr;20(4):366-7. doi: 10.1634/theoncologist.2014-0424. Epub 2015 Mar 16. PMID 25777347
- See also: main page of hadassah hospital - the main facility of this trial — http://WWW.hadassah.org.il